CLINICAL TRIAL: NCT01990989
Title: Clopidogrel Pharmacogenetic Score System Established for Chinese Patients
Brief Title: Clopidogrel Pharmacogenetic Score System
Acronym: CPASS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Tong Yin, Research Associate of Institute of Geriatric Cardiology, Chinese PLA General Hospital
Other Study IDs: 2012042
Record Dates: First submitted 2013-11-18; First posted 2013-11-25 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Acute Coronary Syndrome
Keywords: clopidogrel; pharmacogenomics; CYP2C19; platelet aggregation; score system; ischemic cardiovascular outcomes; hemorrhage complications
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA extracted from peripheral whole blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Clopidogrel treated patients: A consecutive cohort with 500 cases treated with 75mg/day maintenance dose of clopidogrel.

SUMMARY:
The aim of the present study is to evaluate candidate variables,including Cytochrome P450 2C19(CYP2C19) genotypes, clinical and demographic variables,to establish a simple risk score that can be easily adopted by clinicians to identify patients who are at risk for HPR and composite cardiovascular outcomes in Chinese Han patients treated with dual antiplatelet therapy.

DETAILED DESCRIPTION:
There is a large inter-individual variability of biological antiplatelet responsiveness in patients treated with clopidogrel. Our previous study suggested that in clopidogrel treated Chinese patients with acute coronary syndromes(ACS),carriers of at least one CYP2C19 loss-of-function allele could predict greater risk of high on-treatment platelet reactivity (HPR), with the impact mainly attributing to CYP2C19*2. But as we know, CYP2C19*2 could only explain a small proportion of the variability. Various clinical and demographic variables have been considered to influence response to antiplatelet therapy.

Study objectives:

The present study aims to evaluate candidate variables,including CYP2C19 gene polymorphisms, clinical and demographic variables,to establish a simple risk score to identify patients who are at risk for HPR and composite cardiovascular outcomes .

Study design:

Step 1: Population enrollment and medication This mono-center study will be conducted in General Hospital of Chinese People's Liberation Army. Consecutive patients more than 18 years old admitted for ACS will be recruited after giving informed consents. After admission, all enrolled patients will be treated with 100 mg aspirin and 75mg clopidogrel per day. A loading dose of 300 mg clopidogrel will be given to patients undergoing coronary angiography.

Step 2: Clinical and demographic data collection A detailed demographic and medical data will be extracted from medical charts and prescription records. For the development of the risk score system, we will chose variables that are available in routine clinical practice. Clinical candidate variables include smoking history, diabetes,hypertension, renal failure with a serum creatinine>1.5mg/dL-1, hypercholesterolemia, left ventricular dysfunction, age, gender, acute coronary syndrome on admission and co-medication with statins, calcium channel inhibitor, and proton pump inhibitors.

Step 3 : Platelet function measurements and Genotyping After 5 days maintenance dose of clopidogrel administration, blood samples will be drawn for light transmittance aggregometry (LTA) testing, using an APACT-4 aggregometer (LABiTec, Germany). The magnitude of on-treatment platelet reactivity was quantified using LTA with 20µmol/L ADP(adenosine disphosphate) as the agonist. Aggregation was expressed as the maximal percentage change in light transmittance from baseline, with platelet-poor plasma as the reference.

Genomic DNA will be extracted from the peripheral blood leucocytes of each patient. The loss of function alleles, CYP2C19*2 (rs4244285) and CYP2C19*3 (rs4986893), will be genotyped by the polymerase chain reaction(PCR)-ligase detection reactions(LDR)sequencing method.

Step 4: Follow-up At one year, the incidence of composite cardiovascular outcomes will be assessed by review of the patients'charts on re-admission or by telephone interview. Telephone interviewers are blinded with respect to the results of platelet aggregation and genotypes.

Step 5: Statistical analysis and development of risk score Logistic regression and Cox proportional hazards survival regression will be used to develop the risk score system with the candidate variables including clinical and demographic variables, CYP2C19 genotypes, and platelet aggregation.

ELIGIBILITY:
Inclusion criteria:

* Patients more than 18 years old
* Admitted for ACS to the Department of Geriatric Cardiology, General Hospital of Chinese People's Liberation Army
* The diagnosis of ACS according to the American Heart Association/American College of Cardiology (AHA/ACC) criteria, 2012

Exclusion criteria:

* Known contraindication to dual anti-platelet therapy
* History of chronic inflammatory disease
* Steroidal and non-steroidal anti-inflammatory drugs use
* Previous administration of antiplatelet drugs within 1 month before coronary artery angiography
* Illicit drug abuse
* Significant bleeding tendency
* Cerebrovascular events within 3months
* Major surgery within 4 weeks

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: consecutive patients treated with maintenance dose of clopidogrel
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-01 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
high on-treatment platelet reactivity (HPR) | After 30 days maintenance dose of clopidogrel administration
  A threshold of 50% maximal post-procedural aggregation was chosen to define HPR.

SECONDARY OUTCOMES:
Composite ischemia cardiovascular outcomes | 1 year
  The composite of death from cardiovascular causes, non-fatal myocardial infarction, non-fatal stroke , urgent coronal revascularization,and stent thrombosis.
Hemorrhagic complications | 1 year
  The primary clinical safety end point of the study is the 1-year incidence of combined major and minor bleeding events defined according to the Thrombolysis in Myocardial Infarction (TIMI) criteria . TIMI major bleedings include hemoglobin reduction >5 g/dL(with or without obvious bleeding spots) , intracranial hemorrhages, and cardiac tamponade.TIMI minor bleedings include hemoglobin reduction >3 g/dL but ≤5 g/dL ,macroscopic hematuria,hemoptysis,hematemesis,ecchymoma,mucous membrane and other minor bleedings.

CONTACTS AND LOCATIONS:
Overall Officials: Tong Yin, Dr., Principal Investigator — Institute of Geriatric Cardiology, General Hospital of People's Liberation Army, Beijing China
Locations (2):
- China (2):
  - Institute of Geriatric Cardiology, General Hospital of Chinese People's Liberation Army, Beijing, Beijing Municipality
  - Institute of Geriatric Cardiology, Beijing, Beijing Municipality

REFERENCES:
- [Background] Zhang L, Chen Y, Jin Y, Qu F, Li J, Ma C, Yang J, Xu B, Wang H, Li X, Li Y, Zhang Y, Lu C, Yin T. Genetic determinants of high on-treatment platelet reactivity in clopidogrel treated Chinese patients. Thromb Res. 2013 Jul;132(1):81-7. doi: 10.1016/j.thromres.2013.05.006. Epub 2013 May 29. PMID 23726091